CLINICAL TRIAL: NCT05853744
Title: Effect of Aromatherapy on Preoperative Anxiety Level
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Professor, Mongi Slim Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aromatherapy
Record Dates: First submitted 2023-04-29; First posted 2023-05-11 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Anxiety; Aromatherapy; Anesthesia, Spinal; Postoperative Period
MeSH Terms: conditions — Anxiety Disorders | interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sequentially numbered and sealed opaque envelopes method was used to carry out the randomization and allocation.
  These were done by a different doctor from the one caring for the patient in the peri-operative period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C (Experimental): patients receiving aromatherapy using cotton balls impregnated with 3 drops of lavender essential oil inhaled from a distance of 10 cm during 20 minutes and pure oxygen administered through a face mask.
  Interventions: Drug: lavender essential oil inhaled using cotton balls
- Group M (Active Comparator): - Group M: inhaled three drops of lavender oil through a facemask. These three drops were already diluted by five milliliters of distilled water and were sprayed in the area by a nebulizer. A cotton ball soaked with water was put 10 cm next to the patient.
  Interventions: Drug: lavender essential oil inhaled using face mask
- Group P (Placebo Comparator): Placebo group: inhaled five milliliters of distilled water in the same way as the patients in the experimental group and also cotton balls with 3 drops of water are placed near the patient.
  Interventions: Drug: Distilled water

INTERVENTIONS:
Drug: lavender essential oil inhaled using cotton balls — cotton balls impregnated with 3 drops of lavender essential oil inhaled from a distance of 10 cm during 20 minutes and pure oxygen administered through a face mask.
  Other Names: Aromatherapy
  Arms: Group C
Drug: lavender essential oil inhaled using face mask — These three drops were already diluted by five milliliters of distilled water and were sprayed in the area by a nebulizer throughout a face mask. A cotton ball soaked with water was put 10 cm next to the patient.
  Other Names: Aromatherapy
  Arms: Group M
Drug: Distilled water — inhaled five milliliters of distilled water in the same way as the patients in the experimental group and also cotton balls with 3 drops of water are placed near the patient.
  Other Names: Placebo
  Arms: Group P

SUMMARY:
The aim of the study was to evaluate the efficacy of lavender aromatherapy in reducing pre-operative anxiety in patients undergoing surgical procedures under spinal anesthesia.

This was a prospective double blinded randomized controlled trial. After patient's approval, the anxiety level was assessed preoperativetively with Visual Analogue scale-anxiety and APAIS scale. To rule out any lavender sensitivity, all subjects were given a skin patch test. This was accomplished by applying a drop of lavender oil to the back of the hand and covering it with a Tegaderm dressing to prevent inhalation and spread of the oil. After randomisation and allocation, the investigators prooceeded with the intervention preoperatively. In the operating room, the acte under spinal anethesia was performed. Then we collect data postoperatively.

DETAILED DESCRIPTION:
Preoperative anxiety is a common occurrence that has the potential to be harmful, with prevalence rates in the literature ranging from 27% to 80%. Clinical manifestation ranges from malaise to acute stress disorder that meets the criteria of Diagnostic and Statistical Manual of Mental Disorders 5 (DSM5).It is associated with a rise of peri-operative morbidity and mortality. Anti-anxiety medications may be effective but it comes with a number of undesirable adverse effects. Aromatherapy is a non-pharmacological approach that is alluring, affordable, and inexpensive and has minimal side effects, but there aren't enough studies to support its efficacy.

The aim of our study was to evaluate the efficacy of lavender aromatherapy in reducing pre-operative anxiety in patients undergoing surgical procedures under spinal anesthesia.

This was a prospective double blinded randomized controlled trial The patients were seen the night before the surgery, a pre-anesthetic visit was performed.

To rule out any lavender sensitivity, all subjects were given a skin patch test. This was accomplished by applying a drop of lavender oil to the back of the hand and covering it with a Tegaderm dressing to prevent inhalation and spread of the oil.

Surgery day, one hour before operation, vital signs were taken: Heart rate, respiratory rate, pulse oximetry, systolic arterial pressure and diastolic arterial pressure.

Then patients were assessed for anxiety using, Visual Analogue scale-anxiety and APAIS scale.

Next, the investigators proceeded with the intervention and patients were assigned into the 3 group of the study. In the operating room, Spinal anesthesia was performed. After surgery the investigators evaluated anxiety level (VAS-A) and post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* Surgery under spinal anesthesia: continuous or single shot;
* Conscious patient cooperative able to communicate;
* No preoperative cognitive disorder;
* Patient consent;
* American society of anesthesiologists' (ASA) physical status of I-III

Exclusion Criteria:

* Pregnant or breastfeeding women;
* Asthma;
* Chronic obstructive pulmonary disease;
* Allergic to essentials oils;
* Anosmia;
* History of chronic anxiety or depression;
* Neuropsychiatric disorder;
* Use of anti-anxiety medications or anti-depressants;
* Drug addiction;
* Emergency surgery required immediately or within 6 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Anxiety level | before and 30 minutes after the intervention 2 hours befor surgery
  Visual Analogue Scale (minimum value 0 means no anxiety and maximum value 10 means the highest anxiety level)

SECONDARY OUTCOMES:
Pre-operative anxiety and information scale | before and 30 minutes after the intervention 2 hours befor surgery
  Amsterdam anxiety and information scale contains six questions, grouped into two components: anxiety subscale (questions 1, 2, 4, and 5) and the need for information subscale (questions 3 and 6).Questions are scored based on Likert's method from 1 ("not at all") to 5 ("extremely"). For the subscale related to the anxiety, the total score ranges from 4 to 20, while for the part of the scale related to the need for information the range is from 2 to 10. A higher score speaks in favor of a higher level of anxiety and a greater need for information. According to the part of the scale related to preoperative anxiety, a patient with a score ≥11 experiences anxiety; according to the part of the scale related to the need for information related to anesthesia and surgery, patients are classified into those who have little or no need for information (score 2-4), those who have an average (score 5-7) and those who have high information requirements (score 8-10)
Anti-anxiety medications requirement | Fifteen minutes before spinal anesthesia or during the act
  the need of midazolam
Patient satisfaction | 2 hours after the end of the surgery
  Iowa Satisfaction with Anesthesia scale consists of eleven items, which either correspond to positive or negative feelings as follows:
  * Three items aim to assess the patient's pain.
  * Six items investigate the patient's other post-operative sensations.
  * Two items require the patient to record his or her anesthetic experience.
  The offered response for each item is a Likert-like six-point scale, with each response given as a satisfaction score ranging from - 3 to 3:
  * 3 = disagree very much; + 3 = agree very much. Response to" negative" questions are reversed so that, a totally satisfied patient would score +3 on all questions. The total satisfaction score is the unweighted average of these 11 scores, so its expected range is also -3 to +3.

CONTACTS AND LOCATIONS:
Overall Officials: Mhamed Sami MS Mebazaa, Pr, Principal Investigator — Mongi Slim local
Locations (1):
- Mongi Slim hospital, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No